CLINICAL TRIAL: NCT04566848
Title: Determination of Immune Check Point Levels in Paracentesis Samples of Gastrointestinal System Malignancy Cases
Brief Title: The Status of Immune Checkpoints at Gastrointestinal Cancer
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Collaborators: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, M.D. PhD, Istanbul Training and Research Hospital
Other Study IDs: Gastrointestinal checkpoints
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Cancer
Keywords: Pancreatic cancer; Gastric cancer; Colorectal Cancer; Immune checkpoints
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastrointestinal cancers: Patients with advanced stage colorectal cancer, gastric cancer and pancreatic cancer who develop malignant ascites
  Interventions: Diagnostic Test: Flow cytometric analysis
- Control: Patients with intraabdominal ascites with benign reasons (liver cirrhosis, Congestive heart failure, etc.) .
  Interventions: Diagnostic Test: Flow cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow cytometric analysis — Measuring the sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9 levels with flow cytometry

SUMMARY:
Colorectal cancers are the third most common cancer in the world. In advanced stages of colorectal cancers, peritoneal carcinomatosis and intraabdominal acid development occur. Although stomach cancer is the 5th most common cancer in the world, it is the third cancer with the highest mortality. Pancreatic cancer is one of the highest mortality cancers worldwide. Likewise, in advanced stages of stomach and pancreatic cancer, peritoneal carcinomatosis and intra- abdominal acid development occur. It is known that the immune system plays an important role in tumor development or destruction of tumor. Recent studies have shown that tumor cells develop escape mechanisms in the tumor microenvironment to escape from host immunity. It has been reported that differentiation of T cells towards Th2 and regulatory T cells is also effective in tumor progression(6). Changes in the tumor microenvironment and immune checkpoints are important mechanisms that lead to escape from the immune system. Immune checkpoints are on the agenda especially after 2018 Nobel Prize and they are important molecules in revealing the relationship.In our study, it is aimed to evaluate whether there is a difference in immune control points in patients with end-stage colorectal cancer, gastric cancer and pancreatic cancer compared to patients without malignancy, and the relationship of these parameters with patient survival and tumor spread mechanisms.

DETAILED DESCRIPTION:
Colorectal cancers are the third most common cancer in the world. In advanced stages of colorectal cancers, peritoneal carcinomatosis and intraabdominal acid development occur. Although stomach cancer is the 5th most common cancer in the world, it is the third cancer with the highest mortality. Pancreatic cancer is one of the highest mortality cancers worldwide. Likewise, in advanced stages of stomach and pancreatic cancer, peritoneal carcinomatosis and intra- abdominal acid development occur. It is known that the immune system plays an important role in tumor development or destruction of tumor. Recent studies have shown that tumor cells develop escape mechanisms in the tumor microenvironment to escape from host immunity. It has been reported that differentiation of T cells towards Th2 and regulatory T cells is also effective in tumor progression(6). Changes in the tumor microenvironment and immune checkpoints are important mechanisms that lead to escape from the immune system. Immune checkpoints are on the agenda especially after 2018 Nobel Prize and they are important molecules in revealing the relationship.

Programmed Cell Death Protein-1 (PD-1) and its ligand, PD-L1, is an immune control point that acts by blocking T cell receptor signal transduction and co-stimuli. T cell immunoglobulin and mucin domain 3 (TIM-3) are mostly expressed on interferon-gamma-producing T cells, Tregs, dendritic cells, B cells, macrophages, natural killer cells (NK) and mast cells. Enhanced regulation of TIM-3 expression is associated with autoimmune diseases. High TIM-3 expression is associated with suppression of T cell responses and T cell depletion characterized by loss of T cell functions during chronic viral infections and during tumor development. With the clinical success of immune checkpoint inhibitors such as ipilimumab and nivolumab for melanoma and lung cancer, immune checkpoints have received more attention.

The role of the immune system in colorectal cancers has been demonstrated, especially in recent studies, with the effects of tumor-infiltrating lymphocytes (TIL) and immune control points on TILs or immune control point ligands on patient survival. Studies in the literature usually include immunological examinations of patient blood or tumor tissue.

There are many publications in the literature on the study of immunological markers from acid fluid samples for various reasons. In these studies, T and B cell subtypes were examined from acid fluids samples taken from patients with spontaneous ascites, especially ovarian cancer and liver cirrhosis. In the only study conducted on gastrointestinal cancers, immunophenotyping was performed in intraabdominal ascites and blood in 22 advanced gastrointestinal tumor patients, and some cell subgroups were associated with clinical worsening.

In the literature, there is no study on immune control points from intra-abdominal acid fluids specific to gastric and colorectal cancer. In our study, it is aimed to evaluate whether there is a difference in immune control points in patients with end-stage colorectal cancer, gastric cancer and pancreatic cancer compared to patients without malignancy, and the relationship of these parameters with patient survival and tumor spread mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intraabdominal ascites with benign reasons (liver cirrhosis, Congestive heart failure, etc.) for control group
* Patients with advanced stage colorectal cancer, gastric cancer and pancreatic cancer who develop malignant ascites for gastrointestinal cancer group

Exclusion Criteria:

* Pregnant
* Primary immune system failure
* HIV patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intraabdominal ascites with benign reasons (liver cirrhosis, Congestive heart failure, etc.) will be the control group, and patients with advanced stage colorectal cancer, gastric cancer and pancreatic cancer who develop malignant ascites will be the gastrointestinal cancer group
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Immune Checkpoints | 4 months
  sCD25 (IL-2Ra), 4-1BB, B7.2 (CD86), Free Active TGF-β1, CTLA-4, PD-L1, PD-1, Tim-3, LAG-3, Galectin-9

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc. Prof. MD., Principal Investigator — İstanbul Training and Research Hospital; Eyup Kaya, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Istanbul Training and Reseach Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sasidharan Nair V, Toor SM, Taha RZ, Shaath H, Elkord E. DNA methylation and repressive histones in the promoters of PD-1, CTLA-4, TIM-3, LAG-3, TIGIT, PD-L1, and galectin-9 genes in human colorectal cancer. Clin Epigenetics. 2018 Aug 6;10(1):104. doi: 10.1186/s13148-018-0539-3. PMID 30081950
- [Background] Nakano M, Ito M, Tanaka R, Yamaguchi K, Ariyama H, Mitsugi K, Yoshihiro T, Ohmura H, Tsuruta N, Hanamura F, Sagara K, Okumura Y, Nio K, Tsuchihashi K, Arita S, Kusaba H, Akashi K, Baba E. PD-1+ TIM-3+ T cells in malignant ascites predict prognosis of gastrointestinal cancer. Cancer Sci. 2018 Sep;109(9):2986-2992. doi: 10.1111/cas.13723. PMID 30187676
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375